CLINICAL TRIAL: NCT03963453
Title: To Train -or Not to Train? the Role of Physical Exercise As Part of Management in Duchenne Muscular Dystrophy
Brief Title: Regular Physical Exercise in Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Extrastiftelsen (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/260 part II
Record Dates: First submitted 2019-05-09; First posted 2019-05-24 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2021-12

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Physical Therapy Modalities; Exercise; Physical Activity; Exercise Program; Muscular Dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Creatine Kinase (CK level)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Interventional: Regular physical exercise group
  Interventions: Other: Physical Exercise
- Control: Standards of care treatment

INTERVENTIONS:
Other: Physical Exercise — Physical exercise are prescribed to be performed three times per week for a year
  Groups: Interventional

SUMMARY:
This study examine whether an evidence-based individual user-preferred exercise program will increase the physical activity level in boys with Duchenne muscular Dystrophy (DMD).

DETAILED DESCRIPTION:
Regular physical activity is recommended in DMD. However, due to progression of muscle weakness and loss of function, a sedentary lifestyle is normal, and disuse of still functioning muscles leads to a secondary deterioration. Use of steroids have proven to decrease the rate of progression, and also leads to adverse advents like obesity and osteoporosis.

Use of muscle strength training and aerobe exercise in DMD, may optimize muscle function, cardio-respiratory fitness and overall physical activity level, in addition to decrease possible adverse advents.

In this study, children with DMD attending Haukeland University Hospital will be invited to participate (N≈14). The participant's physical activity level is registered during a four week baseline period and follow up. At start, 6 months and 12 months, a five day hospital stay will be conducted, both for testing and to prescribe an individual user preferred physical exercise program. The exercise program will be performed at home between the hospital visits. Benefits, safety and feasibility of regular physical exercise will be examined during follow-up and end of study. For comparison of the physical activity level and motor function, DMD children attending standards of care follow-up at others Norwegian regional pediatric rehabilitation clinics will be invited to participate in a control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with conclusive DMD diagnosis
* Written consent
* Able to perform physical exercise and answer questions

Exclusion Criteria:

* Lack of consent
* Cognitive disabled unable to answer questionnaire, understand instructions, and able to know what they participate in.
* Language difficulties

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — DMD is a X-linked neuromuscular disease
Study Population: Boys with DMD from Hordaland county, attending the pediatric rehabilitation centre at Haukeland university hospital, will be recruited for intervention.
  For comparison, boys with DMD, attending other Norwegian pediatric rehabilitation centres will be invited as control group. Assessment of their physical activity level and self-reported physical activity level will be examined at start and after 12 months. In addition, functional abilities by use of North Star ambulatory assessment or EK2 scale will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | Change from Baseline Physical Activity level at 12 months.
  The participants physical activity level will be monitored by use of an ActiGraph for seven days including a weekend. Two registrations will take place during a four week baseline period, followed by additional registrations at 3, 6, 9 and 12 months (intervention period).

SECONDARY OUTCOMES:
Physical Activity Questionnaire for children (PAQ-C) | Change from Baseline PAQ-C score at 12 months
  The PAQ-C is a self-administrated, 7 day recall instrument, developed to assess general levels of physical activity throughout the elementary school year. The PAQ-C provides a summary physical activity score derived from nine items, each scored on a 5-point scale. The nine items and scores are:
  1. "Spare time activities". Score "no activity" being a 1, "7 times or more" being a 5.
  2. "Physical education". 3. "Recess".4. "Lunch". 5 "Right after school". 6 "Evening". 7 "Weekend". 8. "Describe you best". Each of these 7 item start from lowest activity response (score 1) to the highest activity response (score 5).
  9. How often did you do physical activities for each weekday? None=score 1 Little bit = score 2, Medium = score 3, Often = score 4, Very often = Score 5. Item 9 mean score is reported. Total score 45 represents the participant's general level of physical activity. The participants perform the PAQ-C at baseline and at every hospital visit (start, 6 and 12 months).
Physical Activity Diary | Day 1 (daily for seven days)
  During physical activity registration with use of ActiGraph monitor, the participants and parents are asked to fill out a diary, describing type of physical activity been performed, for how long the physical activity was performed, how tired the participants became, and how did the participant enjoy the activity being performed. In addition the participants is asked to give a summary of the week regarding to name the most enjoyable activity this week and the reason why, and to describe if there occurred something unusual that increased or decreased their physical activity level more than regular.
Pediatric Quality of Life Inventory (PedsQL version 4). Child Report. | Change from Baseline quality of life at 12 months
  The Pediatric Quality of Life Inventory TM (PedsQL TM) is a questionnaire measuring measures quality of life in children, adolescents and young adults. The questionnaire have four subscales with a total of 23 items. Each items with score 0 to 4. The subscales are Physical functioning (eight items), Emotional functioning (five items), Social functioning (five items) and School functioning (five items). A score can be calculated for each subscale. Total score 100 points indicate optimal quality of life. A Psychosocial score can also be calculated (based on the subscales Emotional, Social and School functioning). Participants will report from PedQoL at start and end of study.
North Star Ambulatory Assessment | Change from Baseline functioning at 12 months
  Standardised test for individual with DMD and Spinal Muscular Atrophy able to ambulate. The following physical activities and functions being quantified: Stand, Walk, Stand up from chair, Stand on one leg (right and left), Climb box step (right and left), descend box step (right and left), Get to sitting, Rise from floor, lifts head, Stands on heels, jump, hop on one leg (right and left), run (10 meter timed test). Performed at every three hospital visit during study period.
"Egen Klassification 2- scale" (EK2 scale) | Change from Baseline functioning at 12 months
  Standardised functional assessment for individuals with DMD not able to walk. The following functions and activities are quantified: Ability to use wheelchair, ability to transfer from wheelchair, ability to stand, ability to balance in the wheelchair, ability to move arms, ability to use the hands and arms for eating, ability to turn in bed, ability to cough, ability to speak, physical well-being, Daytime fatigue, head control, ability to control joystick, food textures, eating a meal, swallowing, hand function which of these activities can you do. A total score possible to achieve is 51 points (0-3 point grading on each function), higher score indicating lower degree of functioning. The test will be performed at each hospital visit
Muscular strength- abdominal muscles | Change from Baseline muscular strength at 12 months
  Isometric testing of abdominal muscles. The force being developed will be recorded as Nm and Kg. The participants will be tested at start, after 6 and 12 months.
Muscular strength - hand grip | Change from Baseline muscular strength at 12 months
  Isometric testing of hand grip. The force being developed will be recorded as Nm and Kg. The participants will be tested at start, after 6 and 12 months.
The 6 minutes assisted bicycling test | Change from Baseline physical capacity at 12 months
  Standardized test where participants will perform a 6 minutes arm cycling test, and the distance, heart rate and perceived exhaustion scored at OMNI scale will be recorded. The test will be performed at each of the three hospital visits.
Blood sample - Creatin kinase (CK) value | Day 1, day 3 and day 5.
  Venous blood samples, as biomarker for muscle inflammation or tissue damage, measured by U/L.
  Assessment of CK will be performed for safety reasons due to intervention. Blood samples will be performed three mornings during the hospital visits.
Lung function - Forced Vital Capacity (FVC). | Change from Baseline FVC at 12 months
  Performed by use of spirometry assessment. Measured by liters in absolute value and percent predicted value. Lung function will be measured at each of the three times during study period.
Lung function - Forced Expiratory Flow first second (FEV1). | Change from Baseline FEV1 at 12 months
  Performed by use of spirometry assessment. Measured by liters in absolute value and percent predicted value. Lung function will be measured at each of the three times during study period.
Lung function - FEV1/FVC ratio. | Change from Baseline FEV1/FVC ratio at 12 months.
  Spirometry assessment. The Ratio is calculated in percent value. All participants will be examined at all three hospital visits during study period.
Lung function - Peak Expiratory Flow (PEF). | Change from Baseline PEF at 12 months.
  Spirometry assessment. The maximal airflow achieved during expiration maneuver, measured as liters per second.
Lung function - Slow Vital Capacity (SVC). | Change from Baseline SVC at 12 months
  The Participant's SVC measured as liters / absolute value will be registered at each hospital visit during study period.
Respiratory muscle function - Maximal Inspiratory Pressure (MIP) | Change from Baseline MIP at 12 months
  The Participant's MIP will be measured and registered as absolute value cm water pressure (cm H20) at each hospital visits during the study period.
Respiratory muscle function - Maximal Expiratory Pressure (MEP) | Change from Baseline MEP at 12 months
  The Participant's MEP will be measured and registered as absolute value cm water pressure (cm H20) at each hospital visits during the study period.
Lung function - Peak Cough Flow (PCF) | Change from Baseline PCF at 12 months
  The Participant's PCF will be measured and recorded as absolute value liters per minutes at each hospital visits during the study period.
Body composition - total body fat tissue mass | Change from baseline body fat tissue mass at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify total fat mass (kilogram and percent) at start and end of study period
Body composition - fat tissue mass of the trunk | Change from baseline body fat tissue mass at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify fat mass of the trunk (kilogram and percent) at start and end of study period
Body composition - fat tissue mass of the arms | Change from baseline body fat tissue mass at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify fat mass of the arms (kilogram and percent) at start and end of study period
Body composition - fat tissue mass of the legs | Change from baseline body fat tissue mass at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify fat mass of the legs (kilogram and percent) at start and end of study period
Body composition, Participant's lean tissue mass, total body | Change from baseline body lean tissue mass at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify both total lean tissue mass (kilogram and percent) at start and end of study period
Body composition, Participant's lean tissue mass of the trunk | Change from baseline body lean tissue mass at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify lean tissue mass of the trunk (kilogram and percent) at start and end of study period
Body composition, Participant's lean tissue mass of the arms | Change from baseline body lean tissue mass at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify lean tissue mass of the arms (kilogram and percent) at start and end of study period
Body composition, Participant's lean tissue mass of the legs | Change from baseline body lean tissue mass at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify lean tissue mass of the legs (kilogram and percent) at start and end of study period
Body composition - Bone Mineral Content (BMC), total body | Change from Baseline bone mineral density at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify total BMC (kilogram and percent) at start and end of study period
Body composition - Bone Mineral Content (BMC) of the trunk | Change from Baseline bone mineral density at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify the trunk BMC (kilogram and percent) at start and end of study period
Body composition - Bone Mineral Content (BMC) of the arms | Change from Baseline bone mineral density at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify the arm's BMC (kilogram and percent) at start and end of study period
Body composition - Bone Mineral Content (BMC) of the legs | Change from Baseline bone mineral density at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify the leg's BMC (kilogram and percent) at start and end of study period
Body composition - bone mineral density. Lumbal column | Change from Baseline bone mineral density at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify mineral (grams/ square centimeter) of the lumbar column at start and end of study period.
Body composition - bone mineral density. Hip bone | Change from Baseline bone mineral density at 12 months
  Participants will be assessed using a Lunar iDXA dual x-ray scanner (dxa-scan), to quantify mineral (grams/ square centimeter) of the hip bone at start and end of study period.
Anthropometric measure - age | Day 1
  The participants age measured in years of age will be registered at start and end of study period
Anthropometric measure - body height | Day 1
  The Participant's height measured in centimeter (cm) will be registered at each hospital visit during study period.
Anthropometric measure - body weight | Day 1
  The Participant's body weight measured as kilograms will be measured and registered at each hospital visit during study period
Anthropometric measure - Body Mass Index (BMI) | Day 1
  The Participant's BMI will be calculated by (kg/m2). at each hospital visit during the study period.
Cardiac function - Blood Pressure | Day 2
  The participants systolic and diastolic blood pressure will be registered (mmHg) at start and end of study period
Cardiac function. Echocardiography - Left ventricular mass | Day 2
  Participants will undergo Ultrasound of the heart, using the cube formula indexed by Height (centimeter^2.7), derevid from two dimensional linear left ventricular measurements (gram per meter ^2.7) at start and end of study.
Cardiac function. Echocardiography - Left ventricular (LV) systolic function by ejection fraction | Day 2
  Participants will undergo Ultrasound of the heart, measuring LV ejection fraction (%) derived from 2D linear LV measurements (Teichholz) at start and end of study.
Cardiac function. Echocardiography - Left ventricular (LV) systolic function by biplane Simpson | Day 2
  Participants will undergo Ultrasound of the heart, measuring LV ejection fraction (%) derived from 2D linear LV measurements (Teichholz) at start and end of study.
Cardiac function. Echocardiography - Left ventricular (LV) systolic function by tissue doppler | Day 2
  Participants will undergo Ultrasound of the heart, measuring LV systolic tissue Doppler (meter/second) at start and end of study.
Cardiac function. Echocardiography - Left ventricular (LV) systolic function by speckle tracking | Day 2
  Participants will undergo Ultrasound of the heart, measuring LV global, longitudinal 2D speckle tracking (%) at start and end of study.
Cardiac function. Echocardiography - Left ventricular (LV) diastolic function by tissue doppler | Day 2
  Participants will undergo Ultrasound of the heart, measuring the ratio of doppler transmitral flow (E) and tissue doppler derived early diastolic velocity (E merk) (without any unit) at start and end of study.
Cardiac function. Echocardiography - Left ventricular (LV) diastolic function by isovolumic relaxation time (IVRT) | Day 2
  Participants will undergo Ultrasound of the heart, measuring IVRT in milliseconds (ms) at start and end of study.
Cardiac function. Electro cardiogram (ECG), heart rate (HR) | Day 2
  Participants will undergo ECG, measuring HR beats per minute at start and end of study.
Cardiac function. Electro cardiogram (ECG) - QRS duration | Day 2
  Participants will undergo ECG, measuring QRS by milliseconds at start and end of study.
Cardiac function. Electro cardiogram (ECG) - PR interval | Day 2
  Participants will undergo ECG, measuring PR interval by milliseconds at start and end of study.
Cardiac function. Electro cardiogram (ECG) - QT time | Day 2
  Participants will undergo ECG, measuring PR interval by milliseconds at start and end of study.
Cardiac function. Electro cardiogram (ECG) - QT time corrected | Day 2
  Participants will undergo ECG, measuring QT time corrected by milliseconds at start and end of study.
Cardiac function. Electro cardiogram (ECG) - QRS axis | Day 2
  Participants will undergo ECG, measuring QRS axis in grades at start and end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Matre, PhD, Study Chair — Orthopedic Clinik, Haukeland University Hospital, PB1400, 5021 Bergen/Norway
Locations (1):
- Department of Physiotherapy. Haukeland University Hospital, Bergen, Norway, Norway

IPD SHARING:
Plan to Share IPD: No